CLINICAL TRIAL: NCT05621447
Title: A Mass Balance Study of [14C] TAS-303 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10060080
Record Dates: First submitted 2022-10-30; First posted 2022-11-18 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — TAS-303

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-303, [14C]TAS-303 (Experimental)
  Interventions: Drug: TAS-303, [14C]TAS-303

INTERVENTIONS:
Drug: TAS-303, [14C]TAS-303 — oral administration on day 1

SUMMARY:
To evaluate the pharmacokinetics, mass balance recovery, metabolite profile and metabolite identification of [14C]TAS-303 following oral single dose

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects who provided written informed consent to participate in the study
2. Aged 18 years or older and younger than 40 years at the time of informed consent
3. Capable of oral intake.
4. Body weight of 50 kg or more and body mass index of 18.5 or more and less than 25.0
5. Had blood pressure, pulse rate, and body temperature meeting any of the following at screening:

Systolic blood pressure: ≧90 mmHg and ≦139 mmHg, Diastolic blood pressure: ≧40 mmHg and ≦89 mmHg, Pulse rate: ≧40 beats per minute (bpm) and ≦99 bpm, Body temperature: ≧35.0°C and ≦37.4°C

Exclusion Criteria:

1. Had current or previous hypersensitivity or allergy to drugs
2. Had current or previous drug abuse (including use of illicit drugs) or alcoholism
3. Had any concurrent disease (including symptoms and signs; however, diseases that do not affect evaluations in the study such as asymptomatic pollinosis and wart are excluded)
4. Received a radioisotope-labeled substance or subject to a large quantity of radiation exposure* within 12 months before the first dose of TAS-303.

   * A large quantity of radiation exposure includes continuous X-ray irradiation, computed tomography (CT) scan, gastric barium test, and positron emission tomography (PET) scan, excluding tests with low radiation exposure (e.g., chest, bone, or dental X-ray examination, or X-ray examination before boarding an airplane).
5. Occupationally exposed to radiation within a year before the first dose of TAS-303 (such as operators who are involved in nuclear power or radiation operations).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Concentrations of total radioactivity in blood and plasma | Day1 to 8 and 10,12,14,16,18,20,22
Plasma TAS-303 concentrations | Day1 to 8 and 10,12,14,16,18,20,22
Maximum plasma concentration (Cmax) | Day1 to 8 and 10,12,14,16,18,20,22
Area under the plasma concentration versus time curve (AUC). | Day1 to 8 and 10,12,14,16,18,20,22
Elimination half life (T1/2) | Day1 to 8 and 10,12,14,16,18,20,22
Radioactivity cumulative excretion rate into urine | Day 1 to Day 22
Radioactivity cumulative excretion rate into feces. | Day 1 to Day 22
Radioactivity excretion and excretion rate，cumulative excretion, cumulative excretion rate in all excreta (urine and feces). | Day 1 to Day 22

SECONDARY OUTCOMES:
Adverse events | Day 1 to Day 29
  The number and incidence of Adverse events.
Treatment-related adverse events | Day 1 to Day 29
  The number and incidence of Treatment-related adverse events.
Number of Participants With Abnormal Laboratory Values | Screening period and Day -2, 8, 15, 22, 29
Blood Pressure | Screening period and Day 1, 2, 8, 15, 22, 29
Pulse rate | Screening period and Day 1, 8, 15, 22, 29
Temperature | Screening period and Day 1, 2, 8, 15, 22, 29
QTc interval | Screening period and Day 1, 8, 15, 22, 29
Heart rate | Screening period and Day 1, 8, 15, 22, 29

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- A site selected by Taiho Pharmaceutical Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Data will not be shared according to the Sponsor policy on data sharing. Taiho policy on data sharing may be found at https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html.